CLINICAL TRIAL: NCT06071507
Title: Management of Malignant Gastric Outlet Obstruction Between Surgery and Endoscopy
Acronym: GOOSE
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: European Pancreatic Club (Unknown); The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other)
Responsible Party: Principal Investigator, Giuseppe Vanella, Principal Investigator, IRCCS San Raffaele
Other Study IDs: GOOSE
Record Dates: First submitted 2023-10-01; First posted 2023-10-06 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Gastric Outlet Obstruction; Pancreatic Cancer
Keywords: Enteral stent; Duodenal stent; Gastroenterostomy; EUS; Bypass; LAMS; Gastrojejunostomy
MeSH Terms: conditions — Gastric Outlet Obstruction; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Enteral Stenting: Endoscopic placement of enteral Self-Expandable Metal Stents (SEMS). The procedure implies endoscopic identification of the stricture, placement of a guidewire through the stricture and placement of a SEMS through the stricture under fluoroscopic control.
- EUS-guided Gastrojejunostomy: The procedure implies distention of the jejunal loop and EUS-guided placement of an electrocautery-enhanced (EC) LAMS connecting the stomach to a jejunal loop distal to the stenosis. Any technique for EUS-GE will be allowed, provided that an EC-LAMS >15mm will be used.
- Surgical Gastrojejunostomy: The procedure implies a surgical anastomosis between gastric wall and a jejunal loop. The procedure can be performed either through laparoscopy or open surgery.

SUMMARY:
The aim of this observational study is to compare the outcomes of three different procedures performed for the management of malignant Gastric Outlet Obstruction due to Pancreatic Cancer.

Patients who undergo:

* Surgical gastroenterostomy
* Endoscopic placement of a self-expanding metallic stent
* EUS-guided gastroenterostomy in accordance with standard clinical practice, will be enrolled to evaluate potential differences between the procedures in terms of clinical success, eating experience, chemotherapy tolerance, and nutritional status during follow-up.

Participants will be asked to complete a quality of life questionnaire at baseline and during follow-up; however, no additional procedures will be conducted as a result of participation in the study.

DETAILED DESCRIPTION:
Gastric Outlet Obstruction (GOO) syndrome is a frequent complication of biliopancreatic and gastroduodenal neoplasms and manifests with recurrent vomiting, dehydration and malnutrition, seriously compromising quality of life and the ability to tolerate chemotherapy.

Standard treatment options for GOO are surgical gastroenterostomy (S-GE) or endoscopic placement of a self-expanding metallic stent (ES): surgical treatment achieves better long-term results at the cost of a more invasive procedure. The advances of therapeutic endosonography (EUS) have provided a new possibility to resolve this condition through EUS-guided gastroenterostomy (EUS-GE). The latter involves the creation of a gastroenteric bypass by endoscopically positioning a lumen-apposing metal stent (LAMS). Recent evidence has shown several advantages over previous treatments, in terms of less invasiveness compared to surgery and greater long-term efficacy compared to enteral stenting. However, most of the evidence comes from retrospective protocols and heterogeneous studies that include different neoplasms and clinical courses. Furthermore, the definition of clinical success in the current literature refers to the resolution of the mechanical obstruction of the syndrome, without any in-depth study on the clinical impact of different management strategies in terms of more complex outcomes, such as survival, quality of life, nutritional status and chemotherapy tolerance.

The aim of this study is to prospectively analyze the long-term clinical impact of GOO management strategies in a homogeneous cohort of patients with pancreatic adenocarcinoma (PC) and recent disease diagnosis.

The design of this study is:

* Observational
* Prospective
* Multicentric
* Comparative (3-arms)

No changes to the current clinical practice of the participating centers are foreseen. Each center will candidate the enrolled patient to the procedure that is routinely and currently used in that clinical scenario at their own center. Enrollment in the protocol does not require additional investigations or treatments, except for the administration of quality-of-life questionnaires. Participation in the study implies sharing of information standardly collected during the oncological journey. The prospective follow-up will address clinical efficacy, safety and patient-reported experience, including assessment of the eating experience, chemotherapy tolerance and nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* cyto-/histo-logically confirmed pancreatic cancer
* a maximum of 6 months from pancreatic cancer diagnosis and candidate to active treatment
* stenosis causing gastric outlet obstruction (GOO) due to neoplastic invasion/compression confirmed by radiology or endoscopy extending from the distal one third of the stomach or the duodenum
* patients candidate to either ES or EUS-GE or s-GE

Exclusion Criteria:

* age < 18 years
* patients with benign or indeterminate gastrointestinal stenosis
* patients with malignant GOO (mGOO) from neoplasia other than pancreatic cancer
* candidates to upfront surgical resection or who already received curative pancreatic resection
* patients who already received a treatment for mGOO
* patients receiving an additional procedure for biliary drainage which might increase the risk of adverse events or hamper the assessment of quality of life; biliary drainage will be allowed if performed uneventfully (without adverse events) at least one day (endoscopic drainage) or one month (surgical hepaticojejunostomy) before mGOO treatment;
* patients carrying any percutaneous drainage (such as percutaneous transhepatic biliary drainage or ascites drainage).
* inability or unwillingness to sign the informed consent form (ICF)
* contraindications to any active palliation of the mGOO, or indication to palliation through venting gastrostomy or nasogastric tube placement alone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A homogeneous population of patients with pathologically confirmed Pancreatic Cancer, candidate to palliation of Gastric Outlet Obstruction and active oncological treatment.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Success | 30 days
  A Gastric Outlet Obstruction Scoring System (GOOSS) >/= 2 after the initial intervention, corresponding to the ability to eat at least soft solids

SECONDARY OUTCOMES:
Eating Experience | 3 months
  Mean difference in the Anorexia Cachexia subscale of the Functional Assessment of Anorexia/Cachexia Treatment (FAACT) scale between pre- and post-procedure
Chemotherapy Tolerance | 24 months
  Delay or discontinuation of an intended chemotherapy regimen
Body Mass Index | 6 months
  A numerical value calculated by dividing a person's weight in kilograms by the square of their height in meters
Body Composition | 6 months
  Muscle area calculated using CT scans using dedicated software
Nutritional status | 6 months
  Evaluated through the Prognostic Nutritional Index, using biochemical values stardardly evaluated during chemotherapy

OTHER OUTCOMES:
Technical Success | Day 0
  completion of the intended procedure
Full diet | 3 months
  GOOSS >/= 3, that is the possibility to eat a full diet
Adverse events | 30 days
  Any post-procedural undesirable event requiring an escalation of medical care (additional investigations or treatments, including medical therapy)
Symptoms recurrence | 24 months
  Persistent recurrence of obstructing symptoms (GOOS Score </=1) after a former clinical success (GOOS Score >/=2)
Overall Survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Vanella, MD, Principal Investigator — IRCCS San Raffaele; Gabriele Capurso, MD, Principal Investigator — IRCCS San Raffaele
Locations (5):
- Hôpital la pitié salpêtrière, APHP, Paris, France
- Italy (2):
  - IRCCS San Raffaele Scientific Institute, Milan
  - ISMETT - University of Palermo, Palermo
- São João University Hospital, Porto, Portugal
- Acibadem Maslak Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeurnink SM, Steyerberg EW, van Hooft JE, van Eijck CH, Schwartz MP, Vleggaar FP, Kuipers EJ, Siersema PD; Dutch SUSTENT Study Group. Surgical gastrojejunostomy or endoscopic stent placement for the palliation of malignant gastric outlet obstruction (SUSTENT study): a multicenter randomized trial. Gastrointest Endosc. 2010 Mar;71(3):490-9. doi: 10.1016/j.gie.2009.09.042. Epub 2009 Dec 8. PMID 20003966
- [Background] van Wanrooij RLJ, Vanella G, Bronswijk M, de Gooyer P, Laleman W, van Malenstein H, Mandarino FV, Dell'Anna G, Fockens P, Arcidiacono PG, van der Merwe SW, Voermans RP. Endoscopic ultrasound-guided gastroenterostomy versus duodenal stenting for malignant gastric outlet obstruction: an international, multicenter, propensity score-matched comparison. Endoscopy. 2022 Nov;54(11):1023-1031. doi: 10.1055/a-1782-7568. Epub 2022 Mar 24. PMID 35325931
- [Background] Bronswijk M, Vanella G, van Malenstein H, Laleman W, Jaekers J, Topal B, Daams F, Besselink MG, Arcidiacono PG, Voermans RP, Fockens P, Larghi A, van Wanrooij RLJ, Van der Merwe SW. Laparoscopic versus EUS-guided gastroenterostomy for gastric outlet obstruction: an international multicenter propensity score-matched comparison (with video). Gastrointest Endosc. 2021 Sep;94(3):526-536.e2. doi: 10.1016/j.gie.2021.04.006. Epub 2021 Apr 20. PMID 33852900
- [Background] Boghossian MB, Funari MP, De Moura DTH, McCarty TR, Sagae VMT, Chen YI, Mendieta PJO, Neto FLP, Bernardo WM, Dos Santos MEL, Chaves FT, Khashab MA, de Moura EGH. EUS-guided gastroenterostomy versus duodenal stent placement and surgical gastrojejunostomy for the palliation of malignant gastric outlet obstruction: a systematic review and meta-analysis. Langenbecks Arch Surg. 2021 Sep;406(6):1803-1817. doi: 10.1007/s00423-021-02215-8. Epub 2021 Jun 14. PMID 34121130